CLINICAL TRIAL: NCT06516536
Title: Interventions Based on Mindfulness and Their Influence on the Mental Health and Healthy Lifestyles of University Students.
Brief Title: Mindfulness and Student Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UJAEN.
Record Dates: First submitted 2024-07-17; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: University Students

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CG) (No Intervention): A control group (CG) that will not undergo treatment, which will be evaluated in the pre and post phase of the study.
- Experimental Group (Experimental): In-person MBI: Intervention from Monday to Thursday, carried out in the first 20 minutes of class. Approach to mindfulness meditation, body scanning and simple yoga postures.
  Interventions: Other: MBI (Mindfulness-Based Intervention)

INTERVENTIONS:
Other: MBI (Mindfulness-Based Intervention) — Breath-Focused Meditation Approach (5-7 minutes):
  They will be guided to observe the flow of air in and out of the nose, noting sensations in the abdomen or chest.
  Body scan (7-8 minutes):
  Students will be guided through a careful exploration of their body. You'll start with your toes and slowly work your way toward your head, paying attention to the physical sensations in each part of your body.
  Simple yoga poses (5-7 minutes):
  Students will stand and follow instructions to perform a series of simple poses, such as mountain pose, tree pose, and cat-cow pose.
  Arms: Experimental Group

SUMMARY:
In recent years, there has been growing interest in the well-being and mental health of college students, driven by a significant increase in mental health problems within this population. Several mindfulness interventions, a technique to improve present moment awareness and emotional acceptance, have shown positive results in improving mental health and developing healthy lifestyle habits in this group.

A recent systematic review with meta-analysis (González et al. 2023) indicates that not only the complete standardized 8-week Mindfulness-Based Stress Reduction (MBSR) program but also other Mindfulness-Based Interventions (MBI) are effective. Compared to MBSR, other MBIs require less time commitment, making them more accessible to a larger population and potentially improving program adherence.

In this study, the researchers compare the results of two interventions, one with MBSR (both in-person and virtual) and another with a shorter MBI (in-person) in a sample of 100 university students. Using four different tools as pre- and post-test measures (Healthy Lifestyle Questionnaire [CEVS-2], Mental Health Continuous Form [MHC-SF], Perceived Stress Scale [PSS], and Mood Regulation Skills Questionnaire). emotions [ERSQ] ]), researchers aim to establish the potential degree of health improvement that different mindfulness interventions can have on the health of university students.

ELIGIBILITY:
Inclusion Criteria:

* Individuals enrolled in university education programs.
* Specific age range that fits the typical characteristics of college students (e.g., 18-25 years old).
* Participants who have given informed consent to participate in the study.
* Students who can commit to participating in the intervention sessions and completing the evaluation questionnaires.

Exclusion Criteria:

* Individuals with medical conditions that could interfere with safe participation in mindfulness sessions (e.g., serious cardiovascular conditions, respiratory disorders).
* Students who have significant difficulties in language comprehension or communication that may affect participation and evaluation.
* Students who are currently actively participating in other similar mindfulness programs could be excluded to avoid bias in the results.
* Individuals with diagnoses of unstabilized serious mental disorders who may require more intensive clinical management.
* Students who are unable to commit to scheduled dates and times for interventions and assessments.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Healthy Lifestyle Questionnaire [CEVS-2] | Up to twelve weeks
  The Healthy Lifestyles Questionnaire (CEVS-2) evaluates habits related to physical activity, nutrition, rest, stress management, social relationships and personal hygiene using a 5-point Likert scale. Higher scores indicate better practices in these aspects, while lower scores suggest areas where improvement could be made.
Mental Health Questionnaire [MHC-SF] | Up to twelve weeks
  The Mental Health Questionnaire (MHC-SF) evaluates mental health in different dimensions using a 5-point Likert scale. Higher scores indicate better mental health status in areas such as emotional, social and psychological well-being, while lower scores may indicate areas of concern or need for support.
The Perceived Stress Scale [PSS] | Up to twelve weeks
  Perceived Stress Scale (PSS). This scale is a self-report instrument that evaluates the level of perceived stress during the last month, it consists of 14 items with a response format of a five-point scale (0 = never, 1 = almost never, 2 = occasionally when, 3 = often, 4 = very often). The total score of the PSS is obtained by reversing the scores of items 4, 5, 6, 7, 9, 10 and 13 (in the following sense: 0=4, 1=3, 2=2, 3=1 and 4 =0) and then adding the 14 items. The direct score obtained indicates that a higher score corresponds to a higher level of perceived stress.
Emotional Regulation Questionnaire [ERSQ]) | Up to twelve weeks
  evaluates emotional regulation strategies using a 5-point Likert scale. Higher scores indicate a more effective and healthy use of strategies to manage and regulate emotions, while lower scores may indicate difficulties in this aspect.

CONTACTS AND LOCATIONS:
Locations (1):
- Ana María González Martín, Las Palmas de Gran Canaria, Spain